CLINICAL TRIAL: NCT01657019
Title: A Phase 3, Multicenter, Open-label, 12 Month Extension Safety and Tolerability Study of SPD489 in the Treatment of Adults With Binge Eating Disorder
Brief Title: Open Label Extension in Adults With Binge Eating Disorder (BED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD489-345; 2012-003313-34 (EudraCT Number)
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Lisdexamfetamine Dimesylate

ARMS (1):
- Lisdexamfetamine dimesylate (Experimental)
  Interventions: Drug: Lisdexamfetamine dimesylate

INTERVENTIONS:
Drug: Lisdexamfetamine dimesylate — 50 or 70 mg administered orally, once a day for 52 weeks
  Other Names: Vyvanse; SPD489; LDX

SUMMARY:
To evaluate the safety and tolerability of SPD489 administered as a daily morning dose (50 or 70mg) in the treatment of moderate to severe binge eating disorder (BED) in adults

ELIGIBILITY:
Inclusion criteria:

1. Completion of an antecedent SPD489 BED Double-blind Study
2. Subject meets the following Diagnostic and Statistical Manual of Mental Disorders Fourth Edition - Text Revision (DSM-IV-TR) criteria for a diagnosis of BED
3. Subject has a body mass index (BMI) of > or =18 and < or =45

Exclusion criteria:

1. Subject has concurrent symptoms of bulimia nervosa or anorexia nervosa.
2. Subject is considered a suicide risk or risk to harm others

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 604 (Actual)
Dates: Start 2012-08-21 (Actual); Primary Completion 2014-10-21 (Actual); Study Completion 2014-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (89):
- United States (84):
  - Birmingham Research Group, Birmingham, Alabama
  - Radiant Research, Tucson, Arizona
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Southwestern Research, Inc., Beverly Hills, California
  - TRIMED Clinical Trials, Corona, California
  - Pharmacology Research Institute, Encino, California
  - Scripps Clinical Research Services, La Jolla, California
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Pacific Research Partners, LLC, Oakland, California
  - Excell Research, Inc, Oceanside, California
  - PCSD - Feighner Research, San Diego, California
  - Western Affiliated Research Institute, Inc, Denver, Colorado
  - Radiant Research, Inc, Denver, Colorado
  - Florida Clinical Research, Bradenton, Florida
  - Gulfcoast Clinical Research, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Fidelity Clinical Research, Inc, Lauderhill, Florida
  - Compass Research, LLC, Leesburg, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Scientific Clinical Research, Inc, North Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Atlanta Institute of Medicine and Research, Atlanta, Georgia
  - Neurotrials Research, Inc, Atlanta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - American Medical Research, Inc, Oak Brook, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Deaconess Health Center, Newburgh, Indiana
  - Clinical Trials Technology, Inc, Prairie Village, Kansas
  - Cypress Medical Research Center, LLC, Wichita, Kansas
  - Louisana Research Associates, Inc, New Orleans, Louisiana
  - McLean Hospital, Belmont, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Activmed Practices & Research, Methuen, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Charles Psychiatric Associates-Midwest Research Group, Saint Charles, Missouri
  - Robert Lynne Horne, MD, Las Vegas, Nevada
  - Center for Psychiatry & Behavioral Medicine, Inc, Las Vegas, Nevada
  - Global Medical Institues, LLC, Princeton, New Jersey
  - Pacific Institute for Research & Evaluation, Albuquerque, New Mexico
  - Brooklyn Medical Institute, Brooklyn, New York
  - Comprehensive Clinical Development, Jamaica, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - CNS Clinica, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Radiant Research, Inc, Akron, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - Community Research, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Lindner Center of Hope, Mason, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Psychiatric Partners, Llp, Eugene, Oregon
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Oregon Center for Clinical Research, Inc, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc, Salem, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - The Clinical Trial Center, LLC., Jenkintown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research, Inc, Anderson, South Carolina
  - Radiant Research, Inc, Greer, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutions, Inc (CNS Healthcare), Memphis, Tennessee
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Futuresearch Clinical Trials, Austin, Texas
  - Futuresearch Trials of Dallas, LP, Dallas, Texas
  - Texas Center for Drug Development, Inc, Houston, Texas
  - Psychiatric Medical Associates, Plano, Texas
  - Radiant Research, Inc, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Radiant Research, Inc, Murray, Utah
  - Advanced Research Institute, Ogden, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Neuroscience, Inc, Herndon, Virginia
  - Northwest Clinical Research, Bellevue, Washington
  - Summit Research Network (Seattle) LLC, Seattle, Washington
  - Dean Foundation, Middleton, Wisconsin
- Germany (4):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Ernovis GmbH, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Klinische Forschung Hannover-Mitte, Hanover
- Hospital Infanta Leonor, Madrid, Spain

REFERENCES:
- [Result] Gasior M, Hudson J, Quintero J, Ferreira-Cornwell MC, Radewonuk J, McElroy SL. A Phase 3, Multicenter, Open-Label, 12-Month Extension Safety and Tolerability Trial of Lisdexamfetamine Dimesylate in Adults With Binge Eating Disorder. J Clin Psychopharmacol. 2017 Jun;37(3):315-322. doi: 10.1097/JCP.0000000000000702. PMID 28383364

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label extension study to evaluate the long-term safety of SPD489 in adults aged 18-55 years with binge eating disorder (BED) who completed 1 of 3 antecedent studies, all of which tested SPD489 for BED (SPD489-208, SPD489-343, or SPD489-344).
Groups:
- All Participants: Participants initially received lisdexamfetamine dimesylate, 30 mg administered orally, once daily during the dose optimization phase, regardless of their treatment assignment in the antecedent study. The dose was increased to an optimal dose of either 50 or 70 mg administered orally, once daily. Participants received treatment for a total of 52 weeks, then were followed for 1 week.
Period: Overall Study
Arm/Group | All Participants
Started | 604
Completed | 369
Not Completed | 235
Not completed — Withdrawal by Subject | 65
Not completed — Adverse Event | 55
Not completed — Lost to Follow-up | 48
Not completed — Protocol Violation | 6
Not completed — Lack of Efficacy | 3
Not completed — Other | 58

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set, defined as all participants who took at least 1 dose of investigational product and who had at least 1 post-Visit 0 safety assessment in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 599
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (9.98)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 301
  >/= 40 years | 298
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521
  Male | 78

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) as a Measure of Safety
Time Frame: 52 weeks
Population: The Safety Analysis Set was defined as all participants who took at least 1 dose of investigational product and who had at least 1 post-Visit 0 safety assessment in the study.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 599
percentage of participants
  Any TEAE | 84.5
  Serious TEAEs | 2.8

2. Primary Outcome: Number of Participants With a Positive Response on The Columbia Suicide Severity Rating Scale (C-SSRS)
Description: Suicidality was assessed by using the C-SSRS, a semi-structured interview designed to capture the occurrence, severity, and frequency of suicide-related thoughts and behaviors. The interview and rating for the C-SSRS was completed by a clinician who had been successfully trained by the sponsor or designee. The interview was initiated with 5 (yes/no) questions, presented in ascending order of severity, about suicidal ideation. The most severe type of ideation was rated for frequency, duration, controllability, deterrents, and reason. If the answers to the first 2 ideation questions were "yes," the clinician asked questions 3-5. Active suicidal ideation included any participant who answered "yes" to questions 2-5. If the answers to ideation questions 1 and 2 were "no," then the clinician proceeded to 5 (yes/no) questions that addressed suicidal behavior, which was categorized as actual attempt, interrupted attempt, aborted attempt, preparatory acts or behaviors, and completed suicide.
Time Frame: 53 weeks
Population: The Safety Analysis Set, defined as all participants who took at least 1 dose of investigational product and who had at least 1 post-Visit 0 safety assessment in the study.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 597
participants
  Suicidal behavior | 0
  Active suicidal ideation | 2
  Non-suicidal self-injurious behavior | 3

3. Secondary Outcome: Percentage of Participants With an Improved Response on The Clinical Global Impressions of Improvement (CGI-I) Scale
Description: The CGI rating scales permitted the global evaluation of a participant's condition severity and improvement over time. The CGI-I was performed to rate the improvement of a participant's condition on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse) and included a 'not assessed' option. The responses were dichotomized into 2 categories (improved or not improved). Improved included very much improved and much improved; not improved included minimally improved, no change, minimally worse, much worse, and very much worse. Not assessed and missing values were excluded from the percentage calculation.
Time Frame: Weeks 1, 4, 24, and 52, and end of treatment (either Visit 16 [Week 52] or Early Termination)
Population: The Full Analysis Set, defined as all participants in the Safety Analysis Set who had at least 1 post-Visit 0 clinical experience outcome assessment in this study. The Safety Analysis Set was defined as all participants who took at least 1 dose of investigational product and who had at least 1 post-Visit 0 safety assessment in the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 597
percentage of participants
  Visit 1 (Week 1), n=589 | 53.7 [49.6 to 57.7]
  Visit 4 (Week 4), n=572 | 88.5 [85.8 to 91.1]
  Visit 9 (Week 24), n=466 | 92.7 [90.3 to 95.1]
  Visit 16 (Week 52), n=369 | 95.4 [93.2 to 97.5]
  End of Treatment, n=597 | 89.9 [87.5 to 92.3]

4. Secondary Outcome: Change From Baseline in The Global Score for The Eating Disorder Examination Questionnaire (EDE-Q)
Description: The EDE-Q is a 28-item questionnaire measuring eating pathology and is derived directly from the Eating Disorder Examination Interview. The EDE-Q focuses on the past 28 days to assess the main behavioral (eating and purging) and attitudinal features of eating disorders. The 28 items are rated by the participant on a 7-point scale (ranging from 0 to 6), with higher scores indicating increased pathology. The EDE-Q includes 4 subscales: Restraint, Eating Concern, Weight Concern, and Shape Concern. The global score is the average of all 28 items, with a range of 0 to 6. A negative value indicates a favorable result. The values presented are the mean change from baseline.
Time Frame: Baseline, Weeks 4, 24, and 52, and end of treatment (either Visit 16 [Week 52] or Early Termination)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 597
units on a scale
  Visit 4 (Week 4), n=483 | -1.66 (1.156)
  Visit 9 (Week 24), n=391 | -1.95 (1.271)
  Visit 16 (Week 52), n=314 | -1.95 (1.261)
  End of Treatment, n=503 | -1.90 (1.284)

5. Secondary Outcome: Percentage of Participants With a Response to The EuroQoL Group 5 Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Mobility
Description: The EQ-5D-5L is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is represented by a single item with 5 levels of responses, from poor health to good health. The percentages of participants with various responses to the mobility questionnaire are reported. Percentages are based on all participants in the Full Analysis Set with a valid result at the given visit.
Time Frame: End of Treatment (ET; either Visit 16 [Week 52] or Early Termination)
Population: as for outcome 3
Measure: Number; unit: percentage of participants at ET
Arm/Group | All Participants
Number analyzed (Participants) | 555
percentage of participants at ET
  I have no problems in walking about | 91.2
  I have slight problems in walking about | 6.8
  I have moderate problems in walking about | 1.4
  I have severe problems in walking about | 0.4
  I am unable to walk about | 0.2

6. Secondary Outcome: Percentage of Participants With a Response to The EuroQoL Group 5 Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Self Care
Description: The EQ-5D-5L is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is represented by a single item with 5 levels of responses, from poor health to good health. The percentages of participants with various responses to the self care questionnaire are reported. Percentages are based on all participants in the Full Analysis Set with a valid result at the given visit.
Time Frame: End of Treatment (ET; either Visit 16 [Week 52] or Early Termination)
Population: as for outcome 3
Measure: Number; unit: percentage of participants at ET
Arm/Group | All Participants
Number analyzed (Participants) | 555
percentage of participants at ET
  I have no problems washing or dressing myself | 97.1
  I have slight problems washing or dressing myself | 1.8
  Moderate problems washing or dressing myself | 0.7
  I have severe problems washing or dressing myself | 0.2
  I am unable to wash or dress myself | 0.2

7. Secondary Outcome: Percentage of Participants With a Response to The EuroQoL Group 5 Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Usual Activities
Description: The EQ-5D-5L is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is represented by a single item with 5 levels of responses, from poor health to good health. The percentages of participants with various responses to the usual activities questionnaire are reported. Percentages are based on all participants in the Full Analysis Set with a valid result at the given visit.
Time Frame: End of Treatment (ET; either Visit 16 [Week 52] or Early Termination)
Population: as for outcome 3
Measure: Number; unit: percentage of participants at ET
Arm/Group | All Participants
Number analyzed (Participants) | 555
percentage of participants at ET
  I have no problems doing my usual activities | 88.5
  I have slight problems doing my usual activities | 8.3
  Moderate problems doing my usual activities | 2.2
  I have severe problems doing my usual activities | 0.9
  I am unable to do my usual activities | 0.2

8. Secondary Outcome: Percentage of Participants With a Response to The EuroQoL Group 5 Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Pain and Discomfort
Description: The EQ-5D-5L is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is represented by a single item with 5 levels of responses, from poor health to good health. The percentages of participants with various responses to the pain/discomfort questionnaire are reported. Percentages are based on all participants in the Full Analysis Set with a valid result at the given visit.
Time Frame: End of Treatment (ET; either Visit 16 [Week 52] or Early Termination)
Population: as for outcome 3
Measure: Number; unit: percentage of participants at ET
Arm/Group | All Participants
Number analyzed (Participants) | 555
percentage of participants at ET
  I have no pain or discomfort | 71.2
  I have slight pain or discomfort | 20.9
  I have moderate pain or discomfort | 7.0
  I have severe pain or discomfort | 0.9
  I have extreme pain or discomfort | 0

9. Secondary Outcome: Percentage of Participants With a Response to The EuroQoL Group 5 Dimension 5-Level Self-Report Questionnaire (EQ-5D-5L) For Anxiety or Depression
Description: The EQ-5D-5L is one of the most widely used generic index measures of health-related quality of life. It consists of a 5-item descriptive system that measures 5 dimensions of health, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is represented by a single item with 5 levels of responses, from poor health to good health. The percentages of participants with various responses to the anxiety/depression questionnaire are reported. Percentages are based on all participants in the Full Analysis Set with a valid result at the given visit.
Time Frame: End of Treatment (ET; either Visit 16 [Week 52] or Early Termination)
Population: as for outcome 3
Measure: Number; unit: percentage of participants at ET
Arm/Group | All Participants
Number analyzed (Participants) | 555
percentage of participants at ET
  I am not anxious or depressed | 75.9
  I am slightly anxious or depressed | 18.7
  I am moderately anxious or depressed | 4.5
  I am severely anxious or depressed | 0.9
  I am extremely anxious or depressed | 0

ADVERSE EVENTS:
Description: Adverse events were assessed for the Safety Analysis Set, defined as all participants who took at least 1 dose of investigational product and who had at least 1 post-Visit 0 safety assessment in the study.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 17/599
Other Adverse Events (participants affected / at risk) | 447/599
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=599)
Hip fracture (Injury, poisoning and procedural complications) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Pneumonia (Infections and infestations) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Liver function test abnormal (Investigations) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1
Gastroenteritis viral (Infections and infestations) | 1
Adjustment disorder with anxiety (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Helicobacter infection (Infections and infestations) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Diverticulitis (Infections and infestations) | 1
Chest pain (General disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=599)
Constipation (Gastrointestinal disorders) | 41
Diarrhoea (Gastrointestinal disorders) | 26
Dry mouth (Gastrointestinal disorders) | 163
Nausea (Gastrointestinal disorders) | 41
Toothache (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 15
Fatigue (General disorders) | 28
Feeling jittery (General disorders) | 30
Irritability (General disorders) | 36
Gastroenteritis (Infections and infestations) | 14
Gastroenteritis viral (Infections and infestations) | 18
Influenza (Infections and infestations) | 16
Nasopharyngitis (Infections and infestations) | 53
Sinusitis (Infections and infestations) | 35
Upper respiratory tract infection (Infections and infestations) | 68
Urinary tract infection (Infections and infestations) | 27
Blood pressure increased (Investigations) | 26
Heart rate increased (Investigations) | 15
Weight decreased (Investigations) | 19
Decreased appetite (Metabolism and nutrition disorders) | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 16
Dizziness (Nervous system disorders) | 21
Headache (Nervous system disorders) | 79
Hypoaesthesia (Nervous system disorders) | 15
Paraesthesia (Nervous system disorders) | 14
Anxiety (Psychiatric disorders) | 30
Bruxism (Psychiatric disorders) | 35
Initial insomnia (Psychiatric disorders) | 25
Insomnia (Psychiatric disorders) | 74
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 16
Tachycardia (Cardiac disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.